CLINICAL TRIAL: NCT02879409
Title: Does Glycated Hemoglobin Variability in Type 2 Diabetes Differ Depending on the Diabetes Treatment Threshold Used in the Qatari Population: Implication on Diabetes Complication Risk?
Brief Title: HbA1c Variability in Type II Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Cornell Medical College in Qatar (Other)
Collaborators: Hamad Medical Corporation (Industry); Sidra Medicine (Other); University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-00058; NPRP: 8-315-3-065 (Other Grant/Funding Number: Qatar National Research Fund); 14-00058 (Other: Weill Cornell Medical College in Qatar); 15103/15 (Other: Hamad Medical Corporation)
Record Dates: First submitted 2016-07-13; First posted 2016-08-25 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus Type 2
Keywords: HbA1c variability; Diabetes Mellitus Type 2; Diabetes microvascular complications; Diabetes macrovascular complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Gliclazide; Sitagliptin Phosphate; Liraglutide; Pioglitazone; dapagliflozin; Insulin; Insulin Aspart; Insulin Glargine

STUDY DESIGN:
Masking Description: This is an randomized open label clinical trial.
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Treatment arm 1 (Experimental): 75 Type 2 diabetic patients with a gender balance who will have the intervention if/when their FBG >140mg/dl
  Intervention: intensify treatment until their FBG is <90mg/dl, using whatever treatment is clinically appropriate for them using different interventions (Metformin, Gliclazide, Sitagliptin, Dapagliflozin, Liraglutide, Pioglitazone, human insulin), and only intensify it further if their FPG rises to >140mg/dl again.
  Interventions: Drug: Metformin; Drug: Gliclazide; Drug: Sitagliptin; Drug: Liraglutide; Drug: Pioglitazone; Drug: Dapagliflozin; Drug: human insulin
- Treatment arm 2 (Experimental): 75 Type 2 diabetic patients with a gender balance who will have the intervention if/when their FBG >115mg/dl
  Intervention: intensify treatment until FBG is <=115 mg/dl and intensify further if >115 mg/dl again, using what ever clinical treatment is necessary (Metformin, Gliclazide, Sitagliptin, Dapagliflozin, Liraglutide, Pioglitazone, human insulin).
  Interventions: Drug: Metformin; Drug: Gliclazide; Drug: Sitagliptin; Drug: Liraglutide; Drug: Pioglitazone; Drug: Dapagliflozin; Drug: human insulin

INTERVENTIONS:
Drug: Metformin — Initial: 500 mg once daily; dosage may be increased by 500 mg weekly; maximum dose: 2,000 mg once daily
  Other Names: Glucophage
Drug: Gliclazide — There is no fixed-dosage regimen for the management of diabetes mellitus with gliclazide. Dose will be individualized based on frequent determinations of blood glucose during dose titration and throughout maintenance. The 30 mg modified-release tablet equals the 80 mg immediate-release tablet.
  Immediate-release tablet: Initial: 80 mg twice daily; titrate based on blood glucose levels. Usual dosage range: 80 to 320 mg/day (maximum dose: 320 mg/day); dosage of ≥160 mg should be divided into 2 equal parts for twice-daily administration.
  Modified-release tablet: Initial: 30 mg once daily; titrate in 30 mg increments every 2 weeks based on blood glucose levels. Maximum dose: 120 mg once daily
  Other Names: Diamicron; Diamicron MR
Drug: Sitagliptin — Oral: 100 mg once daily
  Other Names: Januvia
Drug: Liraglutide — SubQ: Initial: 0.6 mg once daily for 1 week; then increase to 1.2 mg once daily; may increase further to 1.8 mg once daily if optimal glycemic response not achieved with 1.2 mg daily.
  Other Names: Victoza
Drug: Pioglitazone — Oral, Monotherapy or combination therapy: 15-30 mg once daily
  Patients with heart failure (NYHA Class I or II): Monotherapy or combination therapy: 15 mg once daily
  Other Names: Actos
Drug: Dapagliflozin — 5mg once daily increasing to 10mg once daily as required
  Other Names: Forxiga; Farxiga
Drug: human insulin — insulin dosage and administration according to physician
  Other Names: novorapid; glargine

SUMMARY:
There are numerous possible reasons why it could be speculated that HbA1c variability may affect complication risk. Of interest are the concepts that both laboratory and clinic evidence suggests that periods of sustained hyperglycemia are 'remembered' (metabolic memory), this in turn is recognized to place patients at greater long-term risk of complications. As such it can be speculated that the detrimental effect of variability in HbA1c may be mediated via the same mechanism as 'metabolic memory' phenomenon.

Aims: To determine whether treatment to one of 2 threshold levels will result in one group of type 2 diabetes patients having the same mean HbA1c but with differing HbA1c variability to that of another and related to markers of oxidative stress, inflammation and microvascular complications. To determine whether a difference in HbA1c variability between the 2 groups will reflect in changes in small nerve fibers assessed with the sensitive method of corneal confocal microscopy and cardiac autonomic function testing. To assess the reproducibility of HbA1c measurement from a whole blood samples initially analyzed and then stored at -80C until the end of the study (2-3 years), as well as storing an aliquot of haemolysate, for reanalysis at the end of the study.

In one arm the investigators will intensify treatment in those with FPG>140mg/dl until their FPG is <90mg/dl, using whatever treatment is clinically appropriate for them, and only intensify it further if their FPG rises to >140mg/dl again. In the other group the investigators will intensify if their FPG is >115 mg/dl until it is <=115 mg/dl and intensify further if >115 mg/dl again. A total of 20 visits within a time frame of 2 and half years will be performed. Visits procedures will include routine biochemistry, eGFR, lipids, fasting glucose, insulin and full blood count, HbA1c, SHBG, hsCRP. EPIC and G-PAQ questionnaires will be collected. Autonomic function testing using deep breathing heart rate variability, and a sensitive measure of small fiber neuropathy using corneal confocal microscopy and a 24 hour urine collection for urinary isoprostanes to measure oxidative stress will be performed, at baseline, 12 and 24 months.

DETAILED DESCRIPTION:
One of the last unanswered question in relation to the influence of glycemic control on diabetes complications is whether increased month-to-month changes in blood glucose (as measured by variability in glycated hemoglobin (HbA1c)) compounds the complication rate and if this can be altered with intervention. Qatar has a high prevalence of diabetes, affecting approximately 23% of the adult population (International Diabetes Federation 2014) that is going to lead to the development of both microvascular and macrovascular complications resulting in the increased morbidity and mortality associated with the disease. The fact that improved glucose control in type 2 as well as type 1 diabetes reduces the risk of microvascular complications is well established. However, more recently it has been demonstrated that the month-to-month variability (the 'rises and falls') in glucose control are also associated with an increased risk of developing these diabetes-associated problems. An individual's long term measure of blood glucose control is represented by the amount of HbA1c measured in the blood. The HbA1c level changes slowly over a much longer period than the constantly fluctuating glucose levels, giving a good indication of overall glucose control in the preceding 2-3 months. What is not known is whether interventions to reduce variability in HbA1c could, in turn, lead to a reduction in diabetes complications. For example even when HbA1c mean is the optimal 7%, there can be high variability in the HbA1c measures (large standard deviation) that may still lead to complications.

This study proposes to gather data to determine whether different treatment thresholds for diabetes in Qatar people have inherently different effects on the variability of HbA1c on a month-to-month basis. By establishing an understanding of how different treatment regimens for hyperglycemia may affect HbA1c variability, this study would then inform on a long term study designed to determine whether interventions to reduce HbA1c variability can reduce micro- or macrovascular complication risk independently of mean HbA1c. If proven, this concept would allow patients to help avoid glycaemia-related vascular complications without having the high potential risk of hypoglycemia that is associated with the current gold standard of diabetes care.

The investigators plan to recruit 150 patients on any glucose lowering medication (HbA1c 7.5-9%), randomize them into one of two treatment threshold groups and test their HbA1c every 6 weeks for 20 visits (visit 1 baseline; therefore 114 weeks) to assess the HbA1c variability of each group. Self-monitored fasting plasma glucose (FPG) measurement will be undertaken 3 times weekly and reported back to the medical team as part of the safety monitoring. Patients will be randomly divided into 2 treatment thresholds. In one the investigators will intensify treatment in those with FPG>140mg/dl until their FPG is <90mg/dl, using whatever treatment is clinically appropriate for them, and only intensify it further if their FPG rises to >140mg/dl again. In the other group Investigators will intensify if their FPG is >115 mg/dl until it is <=115 mg/dl and intensify further if >115 mg/dl again. As such the study will be treatment threshold dependent and therapy independent. This will help circumvent any concern that the drug regimen could complicate the analysis or present a confounder. In practical terms it means the investigators give both groups of patients the same therapy that is intensified according to the treatment threshold with the addition of the same hypoglycemic agents as used in routine clinical practice. Intensifying treatment dose would be undertaken if three consecutive FPG were above the target of 140 or 115 mg/dl. This will be advised by the patient ringing the study coordinator and/or the study coordinator ringing the patient weekly and advising the consultant what the FPG values are for action. It is anticipated that the mean HbA1c will be comparable but the variability of the HbA1c will differ between the 2 populations.

Whole blood samples taken from the recruited patients will be freshly analyzed in a biochemical and HbA1c analyzer. Following this the samples and an aliquot of haemolysate will be stored at -80C for 2-3 years (the duration of the study), when they will be reanalyzed at the completion of the study and the results will be compared with the measurements prior to storage.

All patients entering the study will be assessed by a dietician at Hamad hospital and advised how to complete the food frequency questionnaire that was devised for an Arab population and based on EPIC. It will be completed every six weeks at the time that the HbA1c is taken. Patients will also be asked to fill in the WHO Global Physical Activity Questionnaire (G-PAQ) that has been translated into Arabic and will be collected on a six weekly basis.

Measurement of the serum lipids (total cholesterol, HDL), inflammatory marker (hsCRP) will be undertaken every 6 weeks when the HbA1c is measured. Twenty four hour urinary oxidative stress (urinary isoprostanes by LC/MS) will be measured at baseline, 12 and 24 months. These measures may provide some insight on the mechanism by which HbA1c variability may alter microvascular and macrovascular risk.

Measures for microvascular complications have been included and these include albumin/creatinine ratio and eGFR that will be undertaken every 4 months as a measure for nephropathy. For neuropathy, autonomic function testing using deep breathing heart rate variability, corneal nerve fiber density (CNFD), a sensitive measure of small fiber neuropathy will be performed at baseline, 12 and 24 months under the expertise of Professor Malik who has established the techniques here in Doha.

Recruitment of the patients:

Only Qatari patients will be recruited and the investigators will aim to recruit a gender balance that reflects that of the local eligible diabetes patients until 150 are recruited aged 18-65 years of age. Patients can be on any treatment including insulin as the study is aiming to look at treatment thresholds, rather than actual treatments. This would mean that patients might have additional medication added or substituted in order to reach the necessary threshold of the study. Patients who may be suitable will be given an information sheet detailing the study and asked to contact the designated coordinator within 2 days. After informed consent that will follow"HRP-803 and HRP-802 INVESTIGATOR GUIDANCE - Documentation of Informed Consent", taken by the study coordinator, subjects will be screened against the inclusion and exclusion criteria for eligibility. Should the patient be suitable for inclusion in the study then blood will be withdrawn for HbA1c, routine biochemistry including creatinine, insulin, fasting glucose, fasting lipids, blood for hsCRP and a full blood count at that visit. Urinary albumin/creatinine will also be assessed. Patients would be randomized at that point. Patients will either attend the clinic or have the study coordinator visit their home every 6 weeks to take blood for HbA1c, routine biochemistry including eGFR, lipids, and hsCRP. Urine for urinary isoprostanes will be taken as a measure of oxidative stress. Urinary albumin/creatinine will also be assessed. This will be undertaken for the 20 study visits to assess their HbA1c variability on their two treatment thresholds. A fasting insulin and glucose will be taken at the beginning, at week 60 and at the end of the study as a measure of insulin resistance (HOMA) to determine if there has been a change in insulin resistance over the course of the study. Sex hormone binding globulin (SHBG) as an indirect measure of insulin resistance will also be taken in the event that the fasting bloods cannot be obtained. Assessment of retinopathy by an ophthalmologist and neuropathy will be undertaken at the beginning, mid point and end of the study that fits with current clinical practice. Renal function will be determined every 6 weeks throughout the study by monitoring GFR and measuring urinary albumin/creatinine. Urinary isoprostanes will be measured using LC/MS in a validated assay that is currently in use.

Autonomic function testing using deep breathing heart rate variability, and a sensitive measure of small fiber neuropathy using corneal confocal microscopy to quantify corneal nerve fiber density (CNFD) will be performed at baseline, 12 months and at 24 months (a total of 3 times over the 2 year study period).

Study Visit Schedule

Visit 1:

* Consent, inclusion and exclusion criteria
* Anthropometric measurement
* Baseline bloods: routine biochemistry including eGFR, lipids, fasting glucose, insulin and full blood count, HbA1c, SHBG, hsCRP.
* Urinary measurements. Urinary albumin/creatinine ratio and isoprostane measurement.
* Randomization into one of the two treatment threshold regimes.
* Autonomic function testing using deep breathing heart rate variability and small fiber nerve measurement using corneal confocal microscopy.

Visits 2-10:

Bloods: HbA1c, lipids. Each specimen will be identified and coded as part of the trial. Urinary isoprostanes will be measured in a validated assay that is currently in use.

Visit 11:

Midpoint of the study Anthropometric measurement: Height, Weight, Waist circumference, blood pressure Baseline bloods: routine biochemistry including sGFR, lipids, fasting glucose, insulin and full blood count, HbA1c, SHBG, hsCRP Urinary measurements: urinary albumin/creatinine ratio 24 hour isoprostane measurement, corneal confocal microscopy and autonomic function assessment performed

Visits 12-20:

Bloods: HbA1c, lipids, eGFR, hsCRP. Each specimen will be identified and coded. 24 hour isoprostane measurement, corneal confocal microscopy and autonomic function assessment performed at visit 20.

Autonomic function testing using deep breathing heart rate variability, and a sensitive measure of small fiber neuropathy using corneal confocal microscopy and a 24 hour urine collection for urinary isoprostanes to measure oxidative stress will be performed, these measurements will be performed at baseline, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Qatari subjects only with type 2 diabetes taking any medication.
* HbA1c 7.5-9.0%.
* Body mass index 26-36.
* Age 18 - 65 years of age.
* Recruitment of a gender balance reflecting the local eligible diabetes patients until 150 are recruited.

Exclusion Criteria:

* Patients with anemia or other conditions known to affect the validity of HbA1c measurement e.g. a haemoglobinopathy known to affect the Hamad HbA1c method or renal failure (CKD Stage 5)
* Patients with concurrent illness
* Patients on medication leading to insulin resistance e.g. corticosteroids
* Pregnancy
* Active retinopathy
* Any clinical exclusion for optimal diabetes control
* Hypoglycemic unawareness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2023-10-01 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Determination of the variability of HbA1c (by measurement of standard deviation of HbA1c) between the 2 diabetes treatment thresholds | 24-30 months
  The primary objective of this study is to determine whether treatment to one of 2 threshold levels will result in one group of type 2 diabetes patients having the same mean HbA1c but with differing HbA1c variability to that of another.

SECONDARY OUTCOMES:
Association of the variability of HbA1c (by measurement of standard deviation of HbA1c) to microvascular changes in heart rate variability, corneal nerve fiber density, albumin/creatinine ratio and estimated glomerular filtration rate. | 24-30 months
  Heart rate variability will be measured by ECG changes to deep breathing. Corneal nerve fiber density will be measured by confocal corneal microscopy
Association of the variability of HbA1c (by measurement of standard deviation of HbA1c) to oxidative stress markers measured by urinary isoprostanes and inflammation measured by highly sensitive C-reactive protein. | 24-30 months
  This will be assessed by comparing the results of HbA1c and it's variability every 6 weeks with results of routine biochemistry including eGFR, lipids, SHBG, hsCRP measured on visit one (initial visit), visit 11 (midpoint of the study), and visit 20 (end of the study).
Comparison of HbA1c (percent) for each subject at baseline and following sample storage of 2 years to assess HbA1c measurement stability. | 2-3 years.
  HbA1c will be measured at the time of the sample collection from fresh and haemolysed blood, then the remaining of the samples will be aliquoted and stored in -80 C then remeasured again after short term storage (2-3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Rayaz Malik, MD PhD, Principal Investigator — Weill Cornell Medicine in Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Kilpatrick ES, Rigby AS, Atkin SL. Effect of glucose variability on the long-term risk of microvascular complications in type 1 diabetes. Diabetes Care. 2009 Oct;32(10):1901-3. doi: 10.2337/dc09-0109. Epub 2009 Jun 23. PMID 19549736
- [Background] Siegelaar SE, Kilpatrick ES, Rigby AS, Atkin SL, Hoekstra JB, Devries JH. Glucose variability does not contribute to the development of peripheral and autonomic neuropathy in type 1 diabetes: data from the DCCT. Diabetologia. 2009 Oct;52(10):2229-32. doi: 10.1007/s00125-009-1473-x. Epub 2009 Aug 12. No abstract available. PMID 19672575
- [Background] Kilpatrick ES, Rigby AS, Atkin SL. The effect of glucose variability on the risk of microvascular complications in type 1 diabetes. Diabetes Care. 2006 Jul;29(7):1486-90. doi: 10.2337/dc06-0293. PMID 16801566
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] UK Prospective Diabetes Study Group. Tight blood pressure control and risk of macrovascular and microvascular complications in type 2 diabetes: UKPDS 38. UK Prospective Diabetes Study Group. BMJ. 1998 Sep 12;317(7160):703-13. PMID 9732337
- [Background] ADVANCE Collaborative Group; Patel A, MacMahon S, Chalmers J, Neal B, Billot L, Woodward M, Marre M, Cooper M, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Liu L, Mancia G, Mogensen CE, Pan C, Poulter N, Rodgers A, Williams B, Bompoint S, de Galan BE, Joshi R, Travert F. Intensive blood glucose control and vascular outcomes in patients with type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2560-72. doi: 10.1056/NEJMoa0802987. Epub 2008 Jun 6. PMID 18539916
- [Background] Duckworth W, Abraira C, Moritz T, Reda D, Emanuele N, Reaven PD, Zieve FJ, Marks J, Davis SN, Hayward R, Warren SR, Goldman S, McCarren M, Vitek ME, Henderson WG, Huang GD; VADT Investigators. Glucose control and vascular complications in veterans with type 2 diabetes. N Engl J Med. 2009 Jan 8;360(2):129-39. doi: 10.1056/NEJMoa0808431. Epub 2008 Dec 17. PMID 19092145
- [Background] Home P. Contributions of basal and post-prandial hyperglycaemia to micro- and macrovascular complications in people with type 2 diabetes. Curr Med Res Opin. 2005 Jul;21(7):989-98. doi: 10.1185/030079905x49662. PMID 16004665
- [Background] Raz I, Wilson PW, Strojek K, Kowalska I, Bozikov V, Gitt AK, Jermendy G, Campaigne BN, Kerr L, Milicevic Z, Jacober SJ. Effects of prandial versus fasting glycemia on cardiovascular outcomes in type 2 diabetes: the HEART2D trial. Diabetes Care. 2009 Mar;32(3):381-6. doi: 10.2337/dc08-1671. PMID 19246588
- [Background] Kilpatrick ES, Rigby AS, Atkin SL. Mean blood glucose compared with HbA1c in the prediction of cardiovascular disease in patients with type 1 diabetes. Diabetologia. 2008 Feb;51(2):365-71. doi: 10.1007/s00125-007-0883-x. Epub 2007 Nov 27. PMID 18040661
- [Background] Waden J, Forsblom C, Thorn LM, Gordin D, Saraheimo M, Groop PH; Finnish Diabetic Nephropathy Study Group. A1C variability predicts incident cardiovascular events, microalbuminuria, and overt diabetic nephropathy in patients with type 1 diabetes. Diabetes. 2009 Nov;58(11):2649-55. doi: 10.2337/db09-0693. Epub 2009 Aug 3. PMID 19651819
- [Background] Marcovecchio ML, Tossavainen PH, Dunger DB. Status and rationale of renoprotection studies in adolescents with type 1 diabetes. Pediatr Diabetes. 2009 Aug;10(5):347-55. doi: 10.1111/j.1399-5448.2009.00510.x. Epub 2009 Jun 2. No abstract available. PMID 19496962
- [Background] Sugawara A, Kawai K, Motohashi S, Saito K, Kodama S, Yachi Y, Hirasawa R, Shimano H, Yamazaki K, Sone H. HbA(1c) variability and the development of microalbuminuria in type 2 diabetes: Tsukuba Kawai Diabetes Registry 2. Diabetologia. 2012 Aug;55(8):2128-31. doi: 10.1007/s00125-012-2572-7. Epub 2012 May 12. PMID 22580991
- [Background] Hirakawa Y, Arima H, Zoungas S, Ninomiya T, Cooper M, Hamet P, Mancia G, Poulter N, Harrap S, Woodward M, Chalmers J. Impact of visit-to-visit glycemic variability on the risks of macrovascular and microvascular events and all-cause mortality in type 2 diabetes: the ADVANCE trial. Diabetes Care. 2014 Aug;37(8):2359-65. doi: 10.2337/dc14-0199. Epub 2014 May 8. PMID 24812434
- [Background] Writing Team for the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group. Effect of intensive therapy on the microvascular complications of type 1 diabetes mellitus. JAMA. 2002 May 15;287(19):2563-9. doi: 10.1001/jama.287.19.2563. PMID 12020338
- [Background] Holman RR, Paul SK, Bethel MA, Neil HA, Matthews DR. Long-term follow-up after tight control of blood pressure in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1565-76. doi: 10.1056/NEJMoa0806359. Epub 2008 Sep 10. PMID 18784091
- [Background] Ihnat MA, Thorpe JE, Ceriello A. Hypothesis: the 'metabolic memory', the new challenge of diabetes. Diabet Med. 2007 Jun;24(6):582-6. doi: 10.1111/j.1464-5491.2007.02138.x. Epub 2007 May 8. PMID 17490424
- [Background] Molitch ME, Steffes MW, Cleary PA, Nathan DM. Baseline analysis of renal function in the Diabetes Control and Complications Trial. The Diabetes Control and Complications Trial Research Group [corrected]. Kidney Int. 1993 Mar;43(3):668-74. doi: 10.1038/ki.1993.96. PMID 8455366
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Molyneaux LM, Constantino MI, McGill M, Zilkens R, Yue DK. Better glycaemic control and risk reduction of diabetic complications in Type 2 diabetes: comparison with the DCCT. Diabetes Res Clin Pract. 1998 Nov;42(2):77-83. doi: 10.1016/s0168-8227(98)00095-3. PMID 9886743
- [Background] Dehghan M, Al Hamad N, Yusufali A, Nusrath F, Yusuf S, Merchant AT. Development of a semi-quantitative food frequency questionnaire for use in United Arab Emirates and Kuwait based on local foods. Nutr J. 2005 May 27;4:18. doi: 10.1186/1475-2891-4-18. PMID 15921524
- [Background] Azmi S, Ferdousi M, Petropoulos IN, Ponirakis G, Fadavi H, Tavakoli M, Alam U, Jones W, Marshall A, Jeziorska M, Boulton AJ, Efron N, Malik RA. Corneal confocal microscopy shows an improvement in small-fiber neuropathy in subjects with type 1 diabetes on continuous subcutaneous insulin infusion compared with multiple daily injection. Diabetes Care. 2015 Jan;38(1):e3-4. doi: 10.2337/dc14-1698. No abstract available. PMID 25538321
- [Background] Jayagopal V, Kilpatrick ES, Jennings PE, Holding S, Hepburn DA, Atkin SL. The biological variation of sex hormone-binding globulin in type 2 diabetes: implications for sex hormone-binding globulin as a surrogate marker of insulin resistance. Diabetes Care. 2004 Jan;27(1):278-80. doi: 10.2337/diacare.27.1.278. No abstract available. PMID 14694008
- [Background] Senn S. Testing for baseline balance in clinical trials. Stat Med. 1994 Sep 15;13(17):1715-26. doi: 10.1002/sim.4780131703. PMID 7997705
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Matthews JN, Altman DG, Campbell MJ, Royston P. Analysis of serial measurements in medical research. BMJ. 1990 Jan 27;300(6719):230-5. doi: 10.1136/bmj.300.6719.230. PMID 2106931
- See also: Weill Cornell Biostatistics core — http://qatar-weill.cornell.edu/research/core-facilities/biostatistics